CLINICAL TRIAL: NCT00554749
Title: What Treatment Works for Children With Selective Mutism? A Treatment Pilot Study
Brief Title: What Treatment Works for Children With Selective Mutism?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regionsenter for barn og unges psykiske helse (Other)
Collaborators: Ullevaal University Hospital (Other)
Responsible Party: Hanne Kristensen, MD, PhD, Centre for Child and Adolescent Mental Health, Eastern and Southern Norway
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1.2006.2116; 15968 (Other: Reg. Committee for medical & health research ethics, Norway)
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Results first posted 2010-11-18 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2010-11

CONDITIONS: Selective Mutism
Keywords: Selective mutism; Children; Treatment
MeSH Terms: conditions — Mutism | interventions — Schools

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 Behavioral intervention (Other): Behavioral intervention in all seven subjects Weekly sessions in the home and the kindergarten using defocused communication and stimulus fading interventions
  Interventions: Behavioral: Interventions at home, in the kindergarten/school

INTERVENTIONS:
Behavioral: Interventions at home, in the kindergarten/school — Weekly interventions including behavior techniques (stimulus fading)
  Other Names: Stimulus fading interventions

SUMMARY:
The purpose of this pilot study is to explore the outcome of a manual based treatment for children with Selective Mutism

DETAILED DESCRIPTION:
Objectives:

The main aim of this pilot study is to increase our knowledge on interventions for Selective Mutism (SM), a childhood condition characterized by a persistent lack of speech in specific situations despite the ability to comprehend and use language. A survey on the treatment offered this group in Norway 1997-2000 showed great variations in therapeutic approach and the overall outcome was poor. Correspondent with the notion of SM as a variant of social anxiety, several case studies have described successful treatments using behaviour techniques (BT's) such as stimulus fading and shaping. In addition, the author's clinical experience is that "defocusing in communication" (e.g. regulation of gaze contact; sitting beside instead of in front of the child, avoiding direct questioning, talking about interesting but impersonal topics) represents another important toil in getting the mute child to start talking. However, to date there are no randomized controlled SM treatment studies, and in fact we know little of what works best to help these children. Our research group has developed an assessment- and treatment manual for children with SM.

In this exploring pilot study referred children with SM aged 3-5 years (n=7) will be given an intervention according to the treatment manual. The intervention is conducted at home and in the kindergarten or at school and includes stimulus fading techniques with weekly sessions. Therapists will be members of the research group or local therapist under supervision.

ELIGIBILITY:
Inclusion Criteria:

* Children with a clinical diagnosis of Selective Mutism (SM)

Exclusion Criteria:

* Children with Mental Retardation (IQ<50)
* Children with Pervasive Developmental Disorder (PDD)
* Children with SM in active treatment
* Children with SM on medication
* Children whose parents are non-Norwegian speaking

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Kristensen, Ph.D., Principal Investigator — Centre of child and adolescent mental health, Eastern and Southern Norway
Locations (1):
- Centre for child and adolescent mental health, Eastern and Southern Norway, Oslo, Norway

RESULTS

PARTICIPANT FLOW:
Recruitment Details: November, 2007 to July, 2008.Location: medical clinic
Groups:
- Behavioral: All participants received identical behavioral treatment with no control group.
Period: Overall Study
Arm/Group | Behavioral
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Behavioral
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 4.30 (0.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Region of Enrollment [Number; unit: participants]
  Norway | 7
School speech questionnaire (SSQ) [Mean (Standard Deviation); unit: units on a scale] — SSQ is a teacher-report measure assessing the frequency of the child's speaking behaviour at school. It is a 9-item questionnaire and each item has four possible responses, ranging 0 (never), 1 (seldom), 2 (often) and (3 always). The standard sum score is added up from the six questions(as defined by its author L. Bergman) and then divided by 6 to make up a corresponding factor score ranging from 0-3(worst value=0,best value=3).
  units on a scale | 0.59 (0.51)

OUTCOME MEASURES:

1. Primary Outcome: School Speech Questionnaire (SSQ)
Description: SSQ is a teacher-report measure assessing the frequency of the child's speaking behaviour at school. It is a 9-item questionnaire. Each item has four possible responses, ranging 0 (never), 1 (seldom), 2 (often) and 3 (always). The standard sum score is added up from the six questions (as defined by its author Lindsey Bergman) and then divided by 6 to make up a corresponding factor score ranging from 0-3.(worst value=0 and best value=3)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Behavioral
Number analyzed (Participants) | 7
Units on a scale | 2.68 (0.35)
Statistical Analysis 1: Comparison: Behavioral; Test type: Superiority or Other; p < 0.001, paired t-test; Paired t-test of SSQ at baseline vs at 6 months, degrees of freedom=6. Difference in SSQ is reported; Mean Difference (Net) = 2.09, 95% CI [1.69 to 2.49], Standard Deviation 0.43

2. Secondary Outcome: Number of Children Who Obtained the Different Treatment Modules (Level of Speaking;Level 1 Through to 6)
Description: 6 Predefined treatment goals reflecting speaking levels from 1 through to 6. 1: Speaks to the therapist(T) in a separate room in the kindergarten with parent (P) present. 2: Speaks to T in a separate room without P. 3: Speaks to a teacher in a separate room with T present. 4: Speaks to other teachers in a separate room with T present. 5: Speaks to teachers in some kindergarten settings without T present. 6: Speaks to teachers in all settings in kindergarten without T present. Each child receives one score at end of treatment according to their acquired level (worst value=1, best value =6)
Time Frame: 6 months
Population: All participants analyzed
Measure: Number; unit: participants
Arm/Group | Behavioral
Number analyzed (Participants) | 7
participants
  Level 6 | 6
  Level 5 | 1
  Level 4 | 0
  Level 3 | 0
  Level 2 | 0
  Level 1 | 0

ADVERSE EVENTS:
Arm/Group | Behavioral
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes